CLINICAL TRIAL: NCT02875236
Title: Efficacy and Safety of OctaplasLG Administration vs. Crystalloids (Standard) in Patients With Septic Shock - a Randomized, Controlled, Open-label Investigator-initiated Pilot Trial
Brief Title: Vasculopathic Injury and Plasma as Endothelial Rescue in Septic Shock Trial. VIPER-Sepsis (EudraCT no. 2016-000707-81)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Changing the study design
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Octapharma (Industry)
Responsible Party: Principal Investigator, Thomas Bech Jørgensen, Consultant, Department of Anesthesia and Intensive Care, Bispebjerg Hospital, Principal Investigator., Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Viper Sepsis
Record Dates: First submitted 2016-08-11; First posted 2016-08-23 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Ringer-acetat
  Interventions: Drug: OctaplasLG®
- Intervention (Active Comparator): OctaplasLG®
  Interventions: Drug: Ringer-acetat

INTERVENTIONS:
Drug: OctaplasLG® — OctaplasLG is an donor plasma product pooled from approximately 1000 single donor units. It possesses unique features when compared to standard fresh frozen plasma, such as having standardized concentrations of natural pro- and anti-coagulation factors, a standardized volume as well as being pathogen free. The manufacturing method of OctaplasLG removes immune complexes and cells in several steps of microfiltration in addition to viral, bacterial and prion pathogen inactivation by immune neutralization. OctaplasLG should reduce the "inflammatory hit" on the endothelium, including the glycocalyx, by having standardized levels of coagulation proteins, which can give more sustainable support to the endothelial regeneration as compared to standard fresh frozen plasma.
  Other Names: OctaplasLG
  Arms: Control
Drug: Ringer-acetat — Crystalloid used as standard of care.
  Other Names: Ringer
  Arms: Intervention

SUMMARY:
Efficacy and safety of octaplasLG® administration vs. crystalloids (standard) in patients with septic shock - a randomized, controlled, open-label investigator-initiated pilot trial.

DETAILED DESCRIPTION:
Recently a great interest in the role of the endothelium in the pathophysiology of sepsis has been introduced. The endothelium is coated by a "thick" endothelial glycocalyx protecting it from becoming activated and prevents capillary leakage. The glycocalyx binds approximately 1-1.5 litres of the plasma portion of the circulating blood and regulates the dynamic exchange between the intra -and extravascular space, therefore, functioning both as a barrier and as a mechano transducer. Damage to the glycocalyx is caused by major trauma, major surgery, or ischemia and reperfusion injury, and resulting in vascular leakage. Damage to the endothelium is further augmented by resuscitation of crystalloids and colloids as well as related to bleeding. Thawed fresh frozen plasma may cause a further "inflammatory hit" towards the glycocalyx and endothelium. The degradation of the glycocalyx increases endothelial permeability with edema formation entitled 'the endothelial leakage syndrome', and resulting in the development of hypotension, pulmonary complications, abdominal compartment syndrome, multi-organ failure and death.

The current strategy for maintaining the intravascular volume in patients with acute critical illness focuses on the administration of crystalloids, such as Ringer-Acetate, and natural colloids. Crystalloids, especially, are known to extravasate and cause edema, which is associated with hypoperfusion and compromised vital organ function by the increased tissue pressure that limits oxygen delivery, and ultimately leading to the complications described above. Until recently, synthetic colloids were the preferred choice of fluids for these patients, but a Scandinavian study in patients with severe sepsis and septic shock (6S trial) demonstrated an increased mortality in patients receiving synthetic colloids, thereby, establishing the adverse effect of such a strategy. Consequently, new resuscitation fluids are needed, preferably not only to support the intravascular volume, but also to support and restore the endothelial integrity.

ELIGIBILITY:
Inclusion Criteria:

* Adult intensive care patients AND
* Septic shock requiring infusion of vasopressor/inotropic agents to maintain blood pressure as defined in international guidelines AND
* Consent obtainable from patient or by proxy (independent physicians and/or next of kin)

Exclusion Criteria:

* Documented refusal of blood transfusion OR
* Treatment with GPIIb/IIIa inhibitors < 24h from screening OR
* Withdrawal from active therapy OR
* Previously within 30 days included in a randomised trial, if known at the time of enrolment OR
* Known Immunoglobulin A deficiency with documented antibodies against Immunoglobulin A OR
* Known hypersensitivity to OctaplasLG: the active substance, any of the excipients (Sodium citrate dihydrate, Sodium dihydrogenphosphate dihydrate or Glycine) or residues from the manufacturing process (Tri (N-Butyl) Phosphate (TNBP) and Octoxynol (Triton X-100)) OR
* Known severe deficiencies of protein S OR
* Pregnancy (non-pregnancy confirmed by patient being postmenopausal or having a negative urine-hCG) OR
* Severe cirrhotic hepatic failure with expected need for treatment with terlipressin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-11-08 (Actual); Study Completion 2016-11-08 (Actual)

PRIMARY OUTCOMES:
Microvascular perfusion | 6 hours after inclusion
  Change in microvascular perfusion as evaluated by sidestream darkfield (SDF; MicroVision Medical, Amsterdam, The Netherlands) imaging technique.
Endothelial activation and damage | 6 hours after inclusion
  Change in biomarkers indicative of endothelial activation and damage (soluble E-selectin, syndecan-1, thrombomodulin, soluble VE-cadherin, nucleosomes)

SECONDARY OUTCOMES:
Mortality | From 6 hours until 90 days
  Difference in mortality between patients receiving active treatment (OctaplasLG®) and standard of care (crystalloids)
Length of stay in Intensive Care Unit | through study completion, an average of 1 month
  Length of stay in the Intensive Care Unit
Vasopressors | through study completion, an average of 1 month
  Days on vasopressors
Ventilator | through study completion, an average of 1 month
  Days on ventilator
Bleeding | 1 week
  Bleeding requiring > 2 RBC / day
SAR | 30 days
  Severe adverse reactions, defined as symptomatic thromboembolism
TACO | 30 days
  Transfusion associated circulatory overload
TRALI | 30 days
  Transfusion Related Acute Lung Injury

OTHER OUTCOMES:
SOFA score | 7 days
  Maximal change in SOFA score
AKI | 7 days
  Acute Kidney Injury (AKI) according to RIFLE Criteria
CRRT | 7 days
  Renal replacement therapy as deemed necessary by the attending physician
TEG | 72 hours
  Thrombelastography maximum amplitude (clot strength) in TEG and TEG Functional Fibrinogen (FF)
DIC | 7 days
  Disseminated intravascular coagulation score (DIC)

CONTACTS AND LOCATIONS:
Overall Officials: Per I Johansson, MD, Study Director — University of Copenhagen, Rigshospitalet, Denmark
Locations (1):
- Intensive Care Unit Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
All data from the study will be made public in a peer review journal after last inclusion. But no individual participant data (IPD) will be public.